CLINICAL TRIAL: NCT04832958
Title: The Role of Imaging Guided Surgery to Improve the Detection of Lymph Node Metastases in Prostate Cancer Patients Treated with Radical Prostatectomy and Extended Pelvic Lymph Node Dissection
Brief Title: Imaging Guided Surgery to Improve the Detection of Lymph Node Metastases in Prostate Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Giorgio Gandaglia, MD, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PSMA RGS
Record Dates: First submitted 2021-04-03; First posted 2021-04-06 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
Keywords: radical prostatectomy; lymph node dissection; lymph node invasion
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radioguided surgery (Experimental): * 68Ga-PSMA PET/MRI acquisition
  * 99mTc-PSMA-I&S intravenous injection the day before surgery
  * 99mTc-PSMA-I&S SPECT/CT imaging
  * 99mTc-PSMA-RGS to detect an increased count rate at the level of the nodal stations
  * Robot-assisted ePLND followed by RP
  * 99mTc-PSMA-RGS to detect an increased count rate in the prostatic fossa after removal of the primary tumor
  * Histopathological examination
  * Monitoring of adverse events and perioperative outcomes after surgery
  Interventions: Drug: 99m-TC-PSMA-I&S

INTERVENTIONS:
Drug: 99m-TC-PSMA-I&S — * 99mTc-PSMA-I&S intravenous injection the day before surgery
  * 99mTc-PSMA-I&S SPECT/CT imaging
  * 99mTc-PSMA-RGS to detect an increased count rate at the level of the nodal stations

SUMMARY:
The project aims at assessing the role of radio-guided surgery in the detection of lymph node invasion (LNI) in prostate cancer (PCa) patients undergoing radical prostatectomy (RP) by using an intraoperative gamma probe and a radioactive labelled PSMA ligand (99mTc-PSMA-I&S). We hypothesize that 99mTc-PSMA-I&S radio-guided surgery (99mTc-PSMA-RGS) might assist physicians in the identification of patients with LNI candidate for an extended pelvic lymph node dissection (ePLND). Overall, 100 men with a LNI risk >5% according to the Briganti nomogram will be submitted to 68Ga-PSMA PET/MRI followed by 99mTc-PSMA-RGS and ePLND. The aims are 1) to assess the safety and tolerability of 99mTc-PSMA-I&S; 2) to assess the accuracy of 99mTc-PSMA-RGS in the identification of LNI compared to available clinical tools and to molecular imaging (i.e., 68Ga-PSMA PET/MRI); 3) to assess whether 99mTc-PSMA-RGS would allow for the identification of positive nodes outside the standard ePLND template.

DETAILED DESCRIPTION:
Potential participants will be identified, screened and recruited by the Urologists working at the Department of Urology, IRCCS San Raffaele, Milan, Italy. A total of 100 patients affected by PCa with a risk of LNI >5% according to the Briganti nomogram and planned to receive RARP with an ePLND according to the European Association of Urology (EAU) guidelines will be identified and enrolled in the study.

The patient must personally sign and date the latest approved version of the Informed Consent Form (ICF) before any trial specific procedures are performed.

Written and verbal versions of the Patient Information and Informed Consent will be presented to the participants detailing no less than:

* The exact nature of the trial
* The surgical procedures
* The implications and constraints of the protocol
* The known side effects and any risks involved in taking part
* The clear statement that the participant is free to withdraw from the trial at any time for any reason without prejudice to future care, and with no obligation to give the reason for withdrawal.

The participant will be allowed as much time as wished to consider the information and the opportunity to question the Investigator, their GP or other independent parties to decide whether they will participate in the trial. Written Informed Consent will then be obtained by means of participant dated signature and dated signature of the person who presented and obtained the Informed Consent. The person who obtained the consent must be suitably qualified and experienced, and have been authorized to do so by the Principal Investigator.

A copy of the signed Informed Consent will be given to the participant. The original signed form will be retained at the trial Centre.

A Patient ID number will be assigned to each patient after the ICF signature: this number corresponds to the Progressive Number assigned in chronological order beginning from 001 (i.e. 001, 002, etc.). For instance, the first patient enrolled will receive the following ID Number: 001.

During Visit 1, the following data will be collected:

* Demographics
* Compliance with inclusion/exclusion criteria
* Informed consent
* Previous & concomitant pathologies/previous significant surgeries (including the Charlson Comorbidity Index)
* Previous & concomitant medications
* Prostate cancer characteristics including PSA values, biopsy grade group, clinical stage and the risk of LNI calculated according to the Briganti nomogram [12]
* Vital signs
* Laboratory testing (absolute neutrophil count; platelets; haemoglobin; serum creatinine) The week before surgery patients will undergo a 68Ga-PSMA PET/MRI or PET/CT scan for preoperative staging. Simultaneous PET/MRI will start 60 minutes after the administration of approximately 160MBq of PSMA with the following protocol: localizer MRI scans to define the number of table positions (PET-FOV) to acquire (4-min/table position); specific attenuation correction and anatomical localization MR sequences at each PET-FOV; pelvic mpMRI protocol according to European Society of Urogenital Radiology guidelines. A positive 68Ga-PSMA PET/MRI will be defined as the presence of any uptake at the level of the pelvic and/or retroperitoneal nodes. The results of this procedure will not change the initially planned treatment.

  99mTc-PSMA-I&S will be intravenously injected the day before surgery (day -1). 99mTc-PSMA-I&S will be prepared using a synthesis kit previously described [25]. SPECT/CT imaging will be performed the same day of treatment administration (day -1) to document positive tracer uptake and will serve as quality control for tracer injection and distribution.

All procedures will be performed through a trans-peritoneal approach using the Da Vinci Xi (Intuitive Surgical, Sunnyvale, CA, USA) robotic Surgical System. The patient will be placed in a Trendelenburg position. After incision of the peritoneum, release of the bladder laterally to the endopelvic fascia, the ureter will be localized.

A drop-in gamma probe will be used for in vivo intraoperative measurements to identify metastatic lesions at the level of the internal iliac, external iliac, obturatory and common iliac stations. A positive finding at PSMA-RGS will be defined as the presence of a count rate of at least twice as compared to the background reference (namely, fatty tissue of each patient). All positive lesions (a count rate of at least twice as compared to the background reference) will be excised. Ex vivo gamma measurements will be performed to immediately to confirm the removal of the radioactive lesion or to prompt further search in case of a missing signal. All the removed tissue will be collected separately according to the site of resection.

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* Age between 18 and 80 years
* Biopsy proven PCa with a LNI risk >5% according to the Briganti nomogram
* Planned to receive a RARP with an ePLND
* Able to understand and willing to sign a written informed consent document

Exclusion Criteria:

* Receipt of neoadjuvant therapies
* Inability to complete the imaging examinations according to the prospective protocol
* Evidence of metastatic disease at conventional imaging before surgery
* Evidence of clinical lymphadenopathies at conventional imaging before surgery
* Life expectancy of less than 12 months
* Previous chemotherapy
* Previous brachytherapy or external beam radiotherapy
* Unstable cardiovascular disease
* Congestive Heart Failure (CHF)
* Clinically significant hepatobiliary or renal disease
* History of significant CNS injuries within 6 months
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial
* Medical history of allergic disease or reactions likely to be exacerbated by the IMPs used in this study or by any of the components of the radiotracers (99mTc-PSMA-I&S and 68Ga-PSMA)
* Patients who received an experimental drug in the context of clinical trials within 30 days from the administration of the radiotracers in the current investigation or within 5 half-lives of the experimental drug itself

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Rate of lymph node invasion | 12 weeks
  Rate of LNI observed at final pathology after 99mTc-PSMA-RGS (histopathological evaluation of the lymph nodes)

SECONDARY OUTCOMES:
Side effects | day 0
  Side effects associated with the administration of 99mTC-PSMA-I&S (day 0)
Postoperative complications | day 28 and day 84
  Rate of intraoperative complications associated with 99mTc-PSMA-RGS assessed at visit 2
Nodal invasion outside the template | 12 weeks
  Rate of LNI observed at final pathology in nodes outside the extended nodal dissection template detected only by 99mTc-PSMA-RGS

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gandaglia G, Mazzone E, Stabile A, Pellegrino A, Cucchiara V, Barletta F, Scuderi S, Robesti D, Leni R, Samanes Gajate AM, Picchio M, Gianolli L, Brembilla G, De Cobelli F, van Oosterom MN, van Leeuwen FWB, Montorsi F, Briganti A. Prostate-specific membrane antigen Radioguided Surgery to Detect Nodal Metastases in Primary Prostate Cancer Patients Undergoing Robot-assisted Radical Prostatectomy and Extended Pelvic Lymph Node Dissection: Results of a Planned Interim Analysis of a Prospective Phase 2 Study. Eur Urol. 2022 Oct;82(4):411-418. doi: 10.1016/j.eururo.2022.06.002. Epub 2022 Jul 22. PMID 35879127